CLINICAL TRIAL: NCT03887208
Title: Evaluation the Safety and Efficacy of the Treatment of Scars and Cutis Laxa Syndrome With the Use of Autologous (Fresh and Stored) Stem Cells Isolated From Adipose Tissue.
Brief Title: Therapy of Scars and Cutis Laxa With Autologous Adipose Derived Mesenchymal Stem Cells
Acronym: 2ABC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Timeless Chirurgia Plastyczna-Janusz Jaworowski (Unknown); Melitus sp. z o.o. (Unknown); Polish Stem Cells Bank S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2ABC Therapy; 2016-004110-10 (EudraCT Number); 267976/13/NCBR/2015 (Other Grant/Funding Number: The National Center for Research and Development, Poland); PL008125 (Other: EU tissue establishment code); Z4217 (Other: ISBT128 (Facility Identification Number))
Record Dates: First submitted 2018-10-30; First posted 2019-03-22 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Skin; Scar; Cutis Laxa; Keloid; Cicatrix
Keywords: scar treatment; cutis laxa treatment; stromal vascular fraction; adipose-derived mesenchymal stem cells
MeSH Terms: conditions — Cicatrix; Cutis Laxa; Keloid | interventions — Laser Therapy; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients receive injections of autologous SVF or ADSC cells isolated in the laboratory from adipose tissue.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous adipose derived stem cells (Experimental): Autologous ADSC injection combined with laser therapy of the skin.
  Interventions: Procedure: Laser therapy; Biological: Autologous ADSC injection
- Placebo - Normal saline injection (Placebo Comparator): Normal sline injection combined with laser therapy of the skin.
  Interventions: Procedure: Laser therapy; Procedure: Normal saline injection

INTERVENTIONS:
Procedure: Laser therapy — non-ablative fractional laser therapy of skin
Biological: Autologous ADSC injection — Subcutaneous injection of autologous ADSC
  Arms: Autologous adipose derived stem cells
Procedure: Normal saline injection — Subcutaneous Normal saline injection
  Arms: Placebo - Normal saline injection

SUMMARY:
The aim of this study is to compare clinical outcomes of patients with large scars or Cutis laxa treated with injections of autologous stromal vascular fraction cells (SVF) and adipose-derived mesenchymal stem cells (ADSC).

DETAILED DESCRIPTION:
Patients suffering from cutis laxa senilis and scars (atrophic, hypertrophic, developed due to surgery, trauma, diseases such as acne vulgaris, post-burn scars) will be treated with product containing - human autologous stromal vascular fraction (SVF) cells and human autologous adipose-derived mesenchymal stem cells (ADSC)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years at the time of qualification to the study
2. Signing informed consent form
3. Women / men
4. Scar or cutis laxa

   Scar eligibility conditions:
   * Area:

     * Stomach
     * Limbs
     * Face
     * Back
     * Chest and neck

       * Onset time: over 6 months
       * Scars previously untreated
       * Atrophic and hypertrophic scars
       * Two scars in close location, each from 2 to 6 cm long and a total surface area of 1 sq. cm to 5 sq. cm or single scar
   * Etiology

     * traumatic
     * burns
     * surgical

   Cutis laxa eligibility conditions:
   * Sun discoloration
   * Pigmentation changes
   * Solar stains
   * Pigment changes also called age spots.
   * Erythema
   * Cracked blood vessels
   * Ruby nevus
   * Atrophic changes of the skin and subcutaneous tissue
   * Changes symmetrically present on both hands
5. Without previous aesthetic treatment in this area, previous standard care.
6. Patient's health which allows anesthesia for liposuction.
7. Ready for follow-up visits

Exclusion Criteria:

1. Active cancer (diagnosed during past 5 years), excluding cured nonmelanoma skin cancer or other non-invasive or in situ cancer (eg. cervical cancer)
2. Active chronic infection
3. Chronic use of NSAIDs
4. Taking any anticoagulant by the patient during 1 hour prior to surgery (excluding prophylactic heparin before liposuction).
5. Coagulation disorders in medical history and actual test results out of normal ranges.
6. Skin infections.
7. Allergies to medications used during liposuction (eg. Lidocaine and derivatives).
8. Status post radiotherapy or chemotherapy
9. Any other disease or condition that may change the evaluation of skin condition (eg. autoimmune disease of the connective tissue)
10. Taking the corticosteroid drugs or cytotoxic medications during the past 30 days
11. Allergy to materials of animal origin
12. Diagnosis of diabetes Type I
13. Diagnosis of AIDS, hepatitis B virus (HBV) or hepatitis C virus (HCV) (positive laboratory test result)
14. Hirsutism or a tattoo at the treatment site
15. Insufficient fat tissue for fat donation
16. Scar after removal of cancer.
17. The patient does not qualify to participate in this study in the opinion of the investigator
18. Pregnancy, breast feeding.
19. Photoallergy or using the drugs causing photoallergy.
20. Active herpes
21. Idiopathic keloids
22. Esthetic or medicinal treatments done previously at the treatment site
23. The use of derivatives of vitamin A during 6 months before the treatment
24. Fitzpatrick phototype V and VI
25. Patients with mental disorders or addicted to drugs and/or alcohol.
26. Participation in other clinical study during the past 6 months.
27. Reactive result of serological and viral tests (ie. HIV-1 and 2 (HIV Ag/ Ab)

    * Hepatitis B Virus Infection, - HbsAg and Anti-hepatitis B core antigen (Anti-HBc);
    * Hepatitis C Virus Infection, Anti-HCV;
    * Syphilis specific tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Change in patient's skin condition | 0-27 weeks
  Evaluation of the effectiveness of the method of application of stem cells in the described indications by evaluating the time after which there will be an improvement of 50% in the point evaluation scale of the quality of life of the patient in relation to the baseline values.
  Scale 1: Impact of skin problems on the quality of life. The aim is to assess to what extent skin ailments have affected the patient's life in the last 2 weeks.
  A five-level scale of evaluation (from 'very strong' to 'not applicable') .The "very strong" value means the worst result, while the "not applicable" value is the best result.
Evaluation of skin problems. Assessment of skin related complaints since the last visit. | 0-27 weeks
  Scale 2: A seven-level grading scale (from "0" to "6").The value "0" means the best result, while "6" is the worst result.
The assessment of the scar by the patient. | 0-27 weeks
  Scale 3: Six-point scale (from '1' to '6'). The value "1" means the best result, while "6" is the worst result.

SECONDARY OUTCOMES:
Changes in volume of the skin (USG) | 0-27 weeks
  Changes in the volume of the fat layer at the application site assessed by skin (USG) thickness.
Changes in skin surface morphology (digital imagining) | 0-27 weeks
  Changes in skin surface morphology assessed by digital imaging.
Record of adverse events | 0-27 weeks
  Evaluation of safety of the method of cells' application assessed by adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Noszczyk-Kostrzewa, PhD, Study Chair — Melitus Ltd; Janusz R Jaworowski, PhD, Principal Investigator — Timeless Ltd
Locations (3):
- Poland (3):
  - Laboratory for Cell Research and Application, Medical University of Warsaw, Warsaw
  - Melitus sp. z o.o., Warsaw
  - Timeless Chirurgia Plastyczna Sp. z o. o., Warsaw